CLINICAL TRIAL: NCT06762821
Title: Clinical and Radiographic Outcomes of Single- Versus Multiple-visit Revascularization of Asymptomatic Necrotic Immature Maxillary Permanent Incisors: a 24-month Randomized Clinical Trial
Brief Title: A 24-month Outcomes of Single- Vs Multiple-visit Revascularization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Osama Seif El-Nasr Hussein Gad El-Hak, Lecturer of Pediatric Dentistry, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20241220284
Record Dates: First submitted 2024-12-23; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Necrotic Immature Permanent Incisors
Keywords: single-visit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: biostatistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-visit revascularization (Experimental): Revascularization protocol will be performed in single visit
  Interventions: Procedure: Single-visit revascularization
- multiple-visit revascularization (Active Comparator): Revascularization protocol will be performed in multiple visits
  Interventions: Procedure: Multiple-visit revascularization

INTERVENTIONS:
Procedure: Single-visit revascularization — Revascularization protocol will be performed in single visit
  Arms: Single-visit revascularization
Procedure: Multiple-visit revascularization — Revascularization protocol will be performed in multiple visit
  Arms: multiple-visit revascularization

SUMMARY:
The current randomized clinical trial will be conducted to evaluate the 24-month clinical and radiographic outcomes after revascularization of asymptomatic necrotic immature permanent maxillary incisors using single- or multiple-visit protocol.

ELIGIBILITY:
Inclusion Criteria:

* Compliant healthy patients who had at least one immature maxillary permanent incisor requiring nonsurgical root canal treatment.
* Patients presenting with a diagnosis of pulp necrosis with chronic apical periodontitis confirmed by history, clinical, radiographic and operative examination.
* Patient without previous endodontic treatment in affected tooth.

Exclusion Criteria:

* Patients with systemic conditions (medical, developmental or behavioral) that make routine dental treatment difficult.
* Patients taking medications that can interfere with healing or hemostasis.
* Patients with allergy to local anesthetics
* Children who will not comply to recall program.
* Teeth with extensive loss of coronal tissue that require restoration with a post
* Teeth with internal or external root resorption

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2024-12-21 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants experiencing Pain after treatment | From enrollment to the end of treatment at 24 months
  Zero is equivalent to no pain and 1 indicates presence of pain that necessitate taking pain killer

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University Dental Hospita, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No
Ethical Considerations